CLINICAL TRIAL: NCT02502006
Title: A Double-blind, Placebo-controlled Investigation of Inter-individual Variability in Pharmacologic Response to Non-steroidal Anti-inflammatory Drugs
Brief Title: Variability in Response to Non-steroidal Anti-inflammatory Drugs
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding was not available to complete enrollment
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 820715; 5U54HL117798 (NIH)
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Non-steroidal Anti-inflammatory Drugs; Healthy volunteers; Celecoxib; Naproxen; Prostaglandin; Cyclooxygenase
MeSH Terms: interventions — Celecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose (Experimental): During each treatment phase, subjects will receive celecoxib (200 mg by mouth twice daily), naproxen (500 mg by mouth twice daily), or placebo (twice daily) for 7 days. Subjects will be instructed to take the study medications twice a day (at approximately 8 AM and 8 PM) on an empty stomach with a full glass of water.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Placebo
- Low dose (Experimental): During each treatment phase, subjects will receive celecoxib (100 mg by mouth twice daily), naproxen (250 mg by mouth twice daily), or placebo (twice daily) for 7 days. Subjects will be instructed to take the study medications twice a day (at approximately 8 AM and 8 PM) on an empty stomach with a full glass of water.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib
  Other Names: Celebrex
Drug: Naproxen
  Other Names: Naprosyn
Drug: Placebo

SUMMARY:
This research study will evaluate inter-individual variability in the response to the non-steroidal anti-inflammatory drugs (NSAIDs), celecoxib and naproxen, among healthy adults. It will also investigate what factors, like age, sex, or genetic background, cause this variability.

DETAILED DESCRIPTION:
Non-steroidal anti-inflammatory drugs (NSAIDs) are commonly used for the treatment of inflammatory pain. Pain is a highly subjective experience, and selecting an analgesic regimen that provides optimal pain relief for a specific patient can be challenging. Moreover, patients often express a preference for a particular NSAID, raising the possibility that the efficacy in relieving pain is variable among individuals. However this has never been studied systematically. The clinical decision-making process has been further complicated by the recognition that NSAIDs cause serious thrombotic adverse events in some patients (1). Elucidating the factors that influence an individual patient's risk of cardiovascular complications and the likelihood of analgesic efficacy will enable clinicians to prescribe NSAIDs rationally in order to maximize their therapeutic benefit while minimizing the risk of adverse cardiovascular events.

NSAIDs are a chemically diverse class of therapeutic agents that exert their analgesic and anti-inflammatory effects via inhibition of cyclooxygenase (COX)-1 and/or COX-2, enzymes that catalyze the first committed step in prostaglandin (PG) synthesis. PGs produce a diverse array of biologic effects via activation of prostanoid receptors, and play important roles in a variety of pathologic and homeostatic processes (2). COX-2 is readily induced in response to pro-inflammatory stimuli and has been considered the primary source of inflammatory PGs. In contrast, the production of PGs with homeostatic functions, such as gastric epithelium cytoprotection, has been ascribed to COX-1, which is constitutively expressed in most tissues (2). Consequently, COX-2-selective NSAIDs, including rofecoxib, valdecoxib, and celecoxib, were developed in order to retain the anti-inflammatory and analgesic effects of inhibition of COX-2-derived PG formation, while avoiding the gastrointestinal toxicity of traditional NSAIDs (i.e. aspirin, ibuprofen, naproxen, etc) that inhibit both isoforms. Although fewer gastrointestinal complications were observed in clinical trials, treatment with COX-2-selective NSAIDs increased the risk of serious cardiovascular adverse events, including myocardial infarction, stroke, and heart failure (1,3).

The risk of thrombotic events associated with the use of NSAIDs, particularly those selective for COX-2, is mediated via suppression of COX-2-derived prostacyclin formation in endothelial and vascular smooth muscle cells (4,5). Prostacyclin possesses potent anti-thrombotic and vasodilatory effects, and thus acts as a general inhibitor of platelet activation in vivo (2). Traditional NSAIDs also inhibit COX-2 in the vasculature, but the associated risk of thrombosis is mitigated to some extent by inhibition of formation of thromboxane A2 (TxA2), a COX-1-derived PG released by activated platelets that promotes platelet activation and aggregation (1,3). Thus, the risk of thrombosis for a particular NSAID is dependent upon its relative selectivity for COX-2 over COX-1 (3,6). In addition to their effects on vascular PG production, all NSAIDs inhibit renal PG formation, resulting in sodium retention and hypertension, which may further augment cardiovascular risk (1,3,7).

Currently, it is recommended that NSAIDs be avoided or used only for a limited duration in patients classified as high cardiovascular risk (8). These recommendations are supported by studies demonstrating that even short-term NSAID use increased the incidence of cardiovascular events in patients undergoing coronary artery bypass grafting (9,10) and following a myocardial infarction (11,12). However, long-term treatment with COX-2-selective NSAIDs also increased the incidence of cardiovascular events in patients considered to be at low baseline risk (13,14), consistent with risk transformation due to atherogenesis and indicating traditional cardiovascular risk factors alone are not sufficient to guide therapeutic decisions. Thus, additional studies are necessary to define comprehensively the factors that modify the cardiovascular risk of NSAID use and facilitate the progressive personalization of NSAID therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women greater than 18 years of age who are non-smokers and in good health based on medical history, physical examination, vital signs, and laboratory tests. Volunteers with adequately controlled hypertension and hyperlipidemia (total cholesterol of ≤270 mg/dL) may participate in the study.

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child.
* Subjects who have received an investigational drug or used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening.
* Subjects with any coagulation, bleeding or blood disorders.
* Subjects who are sensitive or allergic to celecoxib (Celebrex) or naproxen (Naprosyn) or their components.
* Subjects who are sensitive or allergic to aspirin or other NSAIDs.
* Subjects with documented history of any gastrointestinal disorders, including bleeding ulcers.
* History of significant cardiovascular disease (including stroke or TIA), renal, hepatic, respiratory (except infections which longer > 6 months prior to screening), immune, endocrine, hematopoietic disorder or neurological disorders.
* History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer resolved by excision, or carcinoma in situ of the cervix adequately treated).
* Has taken any prescription medication other than hormone replacement therapy (including males taking testosterone as a hormone replacement to treat a documented low testosterone level), thyroid replacement hormones, anti-hyperlipidemic agents, or anti-hypertensive medications. Individuals taking other/additional chronic stable medications can be considered on a case-by-case basis for inclusion in the study if agreed upon by judgment of the investigators.
* Has taken NSAIDs or anti-secretory agents (proton pump inhibitors or H2 receptor antagonists) within 14 days prior to study drug administration
* Has ever taken the any anti-platelet or anti-coagulant agents
* Used dietary or herbal supplements containing salicylates, Vitamin E, fish oil, or any other herbal supplements, within 14 days of study drug administration.
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
* Subjects who have had a history of drug or alcohol abuse within the last 6 months.
* Subjects who are unwilling to provide a blood sample for genetic analyses and creation of a lymphoblastoid cell line.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania, Institute for Translational Medicine and Therapeutics; Tilo Grosser, MD, Principal Investigator — University of Pennsylvania, Institute for Translational Medicine and Therapeutics; Katherine N Theken, PharmD, PhD, Principal Investigator — University of Pennsylvania, Institute for Translational Medicine and Therapeutics; Carsten Skarke, MD, Principal Investigator — University of Pennsylvania, Institute for Translational Medicine and Therapeutics
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Theken KN, Ghosh S, Skarke C, Fries S, Lahens NF, Sarantopoulou D, Grant GR, FitzGerald GA, Grosser T. Degree of Cyclooxygenase-2 Inhibition Modulates Blood Pressure Response. Hypertension. 2026 Feb;83(2):e25516. doi: 10.1161/HYPERTENSIONAHA.124.25516. Epub 2025 Dec 29. PMID 41459594
- [Derived] Theken KN, Ghosh S, Skarke C, Fries S, Lahens NF, Sarantopoulou D, Grant GR, FitzGerald GA, Grosser T. Degree of Cyclooxygenase-2 Inhibition Modulates Blood Pressure Response to Celecoxib and Naproxen. medRxiv [Preprint]. 2024 May 31:2024.05.30.24308244. doi: 10.1101/2024.05.30.24308244. PMID 38854091

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: During each treatment phase, subjects received celecoxib (100 mg by mouth twice daily), naproxen (250 mg by mouth twice daily), or placebo (twice daily) for 7 days. Subjects were instructed to take the study medications twice a day (at approximately 8 AM and 8 PM) on an empty stomach with a full glass of water.
Period: Celecoxib
Arm/Group | All Study Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Naproxen
Arm/Group | All Study Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Placebo
Arm/Group | All Study Participants
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Enrollment: During each treatment phase, subjects will receive celecoxib (100 mg by mouth twice daily), naproxen (250 mg by mouth twice daily), or placebo (twice daily) for 7 days. Subjects will be instructed to take the study medications twice a day (at approximately 8 AM and 8 PM) on an empty stomach with a full glass of water.
Arm/Group | Total Enrollment
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 16
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 22.6 (1.9)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 115.3 (8.9)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 69.8 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: COX-1 Activity ex Vivo
Description: COX-1 activity was measured ex vivo using a whole blood assay. Thromboxane A2 serum concentrations were quantified before, and 0.5, 1, 2, 4, 8, and 12 h after treatment and expressed as AUC over the 12 hour dosing interval.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: ng*h/ml
Groups:
- Celecoxib; Naproxen; Placebo: During each treatment phase, subjects received celecoxib (100 mg by mouth twice daily), naproxen (250 mg by mouth twice daily), or placebo (twice daily) for 7 days. Subjects were instructed to take the study medications twice a day (at approximately 8 AM and 8 PM) on an empty stomach with a full glass of water.
Arm/Group | Celecoxib | Naproxen | Placebo
Number analyzed (Participants) | 16 | 16 | 16
ng*h/ml | 2869 (1357) | 115.7 (66.8) | 3135 (1489)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; Test type: Superiority; p < 0.0001, ANOVA

2. Primary Outcome: COX-2 Activity ex Vivo
Description: COX-2 activity was assessed ex vivo using a whole blood assay. Prostaglandin E2 concentrations in LPS-treated plasma were quantified before, and 0.5, 1, 2, 4, 8, and 12 h after treatment and expressed as AUC over the 12 hour dosing interval.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Celecoxib | Naproxen | Placebo
Number analyzed (Participants) | 16 | 16 | 16
ng*h/ml | 87.86 (49.92) | 54.71 (51.37) | 154.1 (83.31)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; Test type: Superiority; p = 0.0004, ANOVA

3. Primary Outcome: COX-1 Activity in Vivo
Description: COX-1 activity was measured in vivo by quantifying the urinary metabolite of thromboxane A2 before, and 1, 2, 4, 8, and 12 h after treatment, normalized to urinary creatinine and expressed as AUC over the 12 hour dosing interval.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: ng*h/mg creatinine
Arm/Group | Celecoxib | Naproxen | Placebo
Number analyzed (Participants) | 16 | 16 | 16
ng*h/mg creatinine | 8.018 (2.488) | 2.907 (2.143) | 9.509 (3.156)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; Test type: Superiority; p < 0.0001, ANOVA

4. Primary Outcome: COX-2 Activity in Vivo
Description: COX-2 activity was measured in vivo by quantifying the urinary metabolite of prostaglandin I2 before, and 1, 2, 4, 8, and 12 h after treatment, normalized to urinary creatinine and expressed as AUC over the 12 hour dosing interval.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: ng*h/mg creatinine
Arm/Group | Celecoxib | Naproxen | Placebo
Number analyzed (Participants) | 16 | 16 | 16
ng*h/mg creatinine | 1.610 (0.3834) | 1.253 (0.8699) | 2.413 (0.8506)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; Test type: Superiority; p = 0.2217, ANOVA

5. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure was measured over 12 hours using an automatic ambulatory blood pressure monitor.
Time Frame: 12 hours
Population: One participant was excluded from blood pressure analysis due to equipment malfunction and incomplete data
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Celecoxib; Naproxen; Placebo: During each treatment phase, subjects will receive celecoxib (100 mg by mouth twice daily), naproxen (250 mg by mouth twice daily), or placebo (twice daily) for 7 days. Subjects will be instructed to take the study medications twice a day (at approximately 8 AM and 8 PM) on an empty stomach with a full glass of water.
Arm/Group | Celecoxib | Naproxen | Placebo
Number analyzed (Participants) | 15 | 15 | 15
mm Hg | 123.0 (10.0) | 127.1 (10.7) | 124.1 (11.2)
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority; p = 0.77, ANOVA — Adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Naproxen vs Placebo; Test type: Superiority; p = 0.18, ANOVA — Adjusted for multiple comparisons

6. Secondary Outcome: Diastolic Blood Pressure
Description: Blood pressure was measured over 12 hours using an automatic ambulatory blood pressure monitor.
Time Frame: 12 hours
Population: One participant was excluded from blood pressure analysis due to equipment malfunction and incomplete data
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Celecoxib | Naproxen | Placebo
Number analyzed (Participants) | 15 | 15 | 15
mm Hg | 74.8 (8.5) | 76.6 (9.3) | 89.7 (8.7)
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority; p = 0.57, ANOVA — Adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Naproxen vs Placebo; Test type: Superiority; p = 0.07, ANOVA — Adjusted for multiple comparisons

7. Secondary Outcome: Mean Arterial Pressure
Description: Blood pressure was measured over 12 hours using an automatic ambulatory blood pressure monitor.
Time Frame: 12 hours
Population: One participant was excluding from blood pressure analysis due to equipment malfunction and incomplete data
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Celecoxib | Naproxen | Placebo
Number analyzed (Participants) | 15 | 15 | 15
mm Hg | 90.4 (8.4) | 92.9 (8.9) | 89.7 (8.7)
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority; p = 0.88, ANOVA — Adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Naproxen vs Placebo; Test type: Superiority; p < 0.05, ANOVA — Adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment through the final study visit, approximately 3 months.
Arm/Group | Celecoxib | Naproxen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-08-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02502006/Prot_SAP_ICF_000.pdf